CLINICAL TRIAL: NCT05490329
Title: A Multidimensional Digital Approach to Address Vaccine Hesitancy and Increase COVID-19 Vaccine Uptake Among African American Young Adults in the South (Tough Talks COVID)
Brief Title: Addressing Vaccine Hesitancy and Increasing COVID-19 Vaccine Uptake Among African American Young Adults in the South
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Lisa Hightow-Weidman, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-1746; R01MD016834 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Vaccine Uptake
Keywords: Vaccine Hesitancy
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (No Intervention): Research staff will provide COVID vaccine materials from the Centers for Disease Control (CDC) to those participants in the Standard of Care (SOC) arm.
- TT-C Intervention (Experimental): Research staff will provide access to the TT-COVID app for one-month, which will provide knowledge about the COVID-19 vaccine, address mis-information, and include multi-media digital stories from study participant's peers.
  Interventions: Behavioral: Tough Talks COVID

INTERVENTIONS:
Behavioral: Tough Talks COVID — Intervention participants will download the TT-C app from the iOS or Google Play store and complete the intervention within one month.
  Arms: TT-C Intervention

SUMMARY:
The study staff will conduct a hybrid type 1 effectiveness implementation 2-arm trail with 360 Black young adults from Alabama, Georgia, and North Carolina. Participants will be randomized to receive the standard of care (control) or the TT-C intervention arm, each with a balance of 180 participants. Primary effectiveness outcome is COVID-19 vaccine uptake define as receipt of any vaccine (primary series or secondary booster). Secondary effectiveness outcomes are vaccine hesitancy, confidence, and knowledge, attitudes, and beliefs. The study staff will also conduct qualitative interviews with a group of purposively selected AA-YA participants (est. n=12-16) and site staff (est. n=6-8) to assess barriers and facilitators to implementation. The hypothesis is that the intervention arm will be more effective than the control arm at increasing vaccine uptake.

DETAILED DESCRIPTION:
The study staff will recruit and enroll 360 AA-YA from communities in Alabama, Georgia, and North Carolina. After collecting informed consent, participants will be randomized using block randomization to the control condition or TT-C (remote), each with a balanced 180 participants (N=360). The standard of care (SOC) control will be the provision of COVID vaccine materials from the CDC.

After screening eligible and agreeing to be contacted, eligible responses will be reviewed individually by study staff to determine authenticity and legitimacy. In addition to eligibility criteria, staff will review bot detection values as well as location based on IP address & latitude/longitude. If determined eligible, staff complete the Verification CRF and REDCap emails the individual with a unique consent form link to complete. Once completed, REDCap sends the baseline survey linked to their unique ID in REDCap.

After the baseline survey is complete, study staff will randomize the participant with the Randomization CRF to either the intervention or control group. Based on the study arm, study staff will either email the participant with the developed SOC materials or email the participant with a unique link to create their account for the TT-C app. If SOC, study staff will compensate the participant $50 for enrolling.

If participant is randomized to intervention arm, they will be prompted to create their account with the provided link, then will be directed to download and login to the TT-C app. Once account creation is confirmed in the administrator portal, study staff will compensate the participant $50 for enrolling.

TT-C arm: Once enrolled, participants will be emailed a unique link to create their TT-C account and instructions on how to download the TT-C (remote) app from the iOS or Google Play store. They will be asked to complete the intervention within one month. Participants will be compensated $50 for completing the baseline and reminded that they will be asked to return in 1 and 3 months for follow-up.

SOC arm: Research staff will provide COVID vaccine materials from the CDC to those participants in the SOC arm. Participants will be compensated $50 for completing the baseline and reminded that they will be asked to complete 1 and 3-month follow- up surveys. To provide the maximum benefit through this trial, after the completion of the data collection associated with the primary RCT, those randomized to the control arm who still report VH will be offered the opportunity to accept the TT-C intervention delivered remotely.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American/Black
* Able to speak and read English
* Has access to personal smartphone
* Current resident of AL, GA, NC

Exclusion Criteria:

* Aged younger than 18 year or older than 29 years
* Does not identify as African American/Black
* Non-English speaking
* Does not live in Al, GA, NC
* Unable to provide informed consent
* Receipt of full COVID vaccine series (including vaccination and booster or prior participation in a vaccine trial)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hightow-Weidman, MD, MPH, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The results will be shared beginning 9 to 36 months following publication.
Access Criteria: Requesting investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Budhwani H, Stoner MCD, Stocks JB, Browne E, Soberano Z, Bond CL, Michaels J, Mancuso N, Larsen MA, Maragh-Bass AC, Tolley EE, Comello MLG, Muessig KE, Pettifor AE, Hightow-Weidman LB. Tough talks COVID-19 (TT-C) digital health intervention: multistate randomized controlled trial. Sci Rep. 2025 Jul 1;15(1):21988. doi: 10.1038/s41598-025-05386-2. PMID 40594178
- [Derived] Budhwani H, Yigit I, Stocks JB, Stoner MCD, Browne E, Pettifor AE, Hightow-Weidman LB. Development and validation of the mpox stigma scale (MSS) and mpox knowledge scale (MKS). BMC Public Health. 2024 Sep 10;24(1):2469. doi: 10.1186/s12889-024-19868-x. PMID 39256711
- [Derived] Budhwani H, Maragh-Bass AC, Tolley EE, Comello MLG, Stoner MCD, Adams Larsen M, Brambilla D, Muessig KE, Pettifor A, Bond CL, Toval C, Hightow-Weidman LB. Tough Talks COVID-19 Digital Health Intervention for Vaccine Hesitancy Among Black Young Adults: Protocol for a Hybrid Type 1 Effectiveness Implementation Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 13;12:e41240. doi: 10.2196/41240. PMID 36689557

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (Control): Research staff will provide COVID vaccine materials from the Centers for Disease Control (CDC) to those participants in the Standard of Care (SOC) arm.
  To provide the maximum benefit through this trial, after the completion of the data collection associated with the primary RCT, those randomized to the control arm who still report vaccine hesitancy will be offered the opportunity to accept the TT-C intervention delivered remotely. These participants will be asked to use the app for one month and complete follow-up surveys at their 4- and 6-month time points (same surveys used for 1 and 3M). These participants will be compensated for survey completion.
Period: 2-Arm Randomized Control Trial
Arm/Group | Standard of Care (Control) | TT-C Intervention
Started | 180 | 180
Month 1 Survey | 174 | 159
Month 3 Survey | 172 | 154
Completed | 172 | 154
Not Completed | 8 | 26
Not completed — Lost to Follow-up | 8 | 25
Not completed — Withdrawal by Subject | 0 | 1
Period: Standard of Care - App Access Crossover
Arm/Group | Standard of Care (Control) | TT-C Intervention
Started | 129 | 0
Month 4 Survey | 124 | 0
Month 6 Survey | 120 | 0
Completed | 120 | 0
Not Completed | 9 | 0
Not completed — Lost to Follow-up | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Control) | TT-C Intervention | Total
Number analyzed (Participants) | 180 | 180 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 180 | 360
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (3.4) | 23.7 (3.5) | 23.7 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 150 | 299
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 172 | 172 | 344
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 180 | 180 | 360
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 180 | 180 | 360
State of Residence [Count of Participants; unit: Participants]
  Alabama | 34 | 33 | 67
  Georgia | 80 | 80 | 160
  North Carolina | 66 | 67 | 133

OUTCOME MEASURES:

1. Primary Outcome: COVID Vaccine Uptake at Month 1
Description: COVID Vaccine Uptake is measured by changes in self-reported receipt of any primary series or booster vaccination
Time Frame: Month 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Control) | TT-C Intervention
Number analyzed (Participants) | 175 | 164
Participants | 6 | 5

2. Primary Outcome: COVID Vaccine Uptake at Month 3
Description: COVID Vaccine Uptake is measured by changes in self-reported receipt of any primary series or booster vaccination
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Control) | TT-C Intervention
Number analyzed (Participants) | 172 | 154
Participants | 8 | 13

3. Secondary Outcome: COVID Vaccine Confidence
Description: COVID Vaccine Confidence is measured by self-reported ability to receive any primary series of booster vaccination at 1 and 3-month follow-up
  Vaccine confidence was a mean score of 7 items with response options ranging from 1-5, and higher scores indicating greater confidence (5=Strongly Agree). Example items were "vaccines are safe" and "vaccines do a good job in preventing the diseases they are intended to prevent."
  Gilkey MB, Reiter PL, Magnus BE, McRee A-L, Dempsey AF, Brewer NT. Validation of the Vaccination Confidence Scale: A Brief Measure to Identify Parents at Risk for Refusing Adolescent Vaccines. Academic Pediatrics. 2016/01/01/ 2016;16(1):42-49. doi:https://doi.org/10.1016/j.acap.2015.06.007
Time Frame: Up to 3 Months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care (Control) | TT-C Intervention
Number analyzed (Participants) | 172 | 152
score on a scale | 3.57 [3.07 to 4.21] | 3.71 [3.36 to 4.29]

4. Secondary Outcome: COVID Vaccine Hesitancy
Description: COVID Vaccine Hesitancy is measured by self-reported refusal to receive any primary series or booster vaccination at 1 and 3-month follow-up
  Vaccine hesitancy was a mean score of a 9-item scale with response ranging from 1-5, and higher scores indicating greater hesitancy (5=Strongly Disagree). Example items included "vaccines are important for my health" and "vaccines are effective."
  Shapiro GK, Tatar O, Dube E, et al. The vaccine hesitancy scale: Psychometric properties and validation. Vaccine. 2018/01/29/ 2018;36(5):660-667. doi:https://doi.org/10.1016/j.vaccine.2017.12.043
Time Frame: Up to 3 Months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard of Care (Control) | TT-C Intervention
Number analyzed (Participants) | 169 | 150
score on a scale | 2.22 [1.78 to 2.67] | 2.00 [1.56 to 2.56]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the time participants were enrolled. Intervention participants for 3 months; Standard of Care (Control) for 3 or 6 months depending on if they received the app later on.
Arm/Group | Standard of Care (Control) | TT-C Intervention
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT05490329/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT05490329/ICF_001.pdf